CLINICAL TRIAL: NCT05560789
Title: The Effect of Physical Activity in Individuals With Post-bariatric Hypoglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00000190
Record Dates: First submitted 2022-09-19; First posted 2022-09-29 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Hypoglycemia; Roux-en-Y Gastric Bypass; Post-bariatric Hypoglycemia; Physical Activity
Keywords: Post-bariatric hypoglycemia; Exercise; Physical activity; Hypoglycemia; Bariatric surgery
MeSH Terms: conditions — Hypoglycemia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study will assess glucose and hormone responses (insulin, glucagon, GLP-1) during structured exercise on a stationary bicycle ergometer or on a treadmill, up to a duration of 60 minutes, in individuals with a history of post-bariatric hypoglycemia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with Post-bariatric Hypoglycemia Performing Structured Physical Activity (Experimental): Individuals with a confirmed diagnosis of post-bariatric hypoglycemia will perform structured physical activity by cycling on a stationary bicycle ergometer or on a treadmill.
  Interventions: Behavioral: Physical activity (cycling on a stationary bicycle ergometer or walking on a treadmill)

INTERVENTIONS:
Behavioral: Physical activity (cycling on a stationary bicycle ergometer or walking on a treadmill) — At time 0, exercise will be initiated and intensity will be increased at 2 minute intervals to achieve low intensity for 30 minutes (as defined by heart rate target 50-55% of maximum heart rate determined as 220-age). Next, intensity will be increased at 2 minute intervals until the heart rate target for moderate intensity exercise is achieved (55-65% of max heart rate), or the total duration of exercise of up to 60 minutes is achieved.

SUMMARY:
The goal of this pilot study is to evaluate the magnitude of changes in glucose and hormone levels in response to structured exercise in the fasting state in individuals with post-bariatric hypoglycemia (PBH).

This pilot study will assess the adequacy of a protocol to test the following hypotheses: (1) hypoglycemia will develop in individuals with PBH in response to exercise; (2) counterregulatory hormonal responses to hypoglycemia during exercise are impaired in individuals with PBH.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females diagnosed with ongoing post-bariatric hypoglycemia with prior episodes of neuroglycopenia, unresponsive to dietary intervention (low glycemic index, controlled carbohydrate portions) and trial of acarbose therapy at the maximally tolerated dose.
2. Age 18-60 years of age, inclusive, at screening.
3. Willingness to provide informed consent and follow all study procedures, including attending all scheduled visits.

Exclusion Criteria:

Initial general screening will be performed during an initial phone or in person visit (e.g. during a clinical visit). Individuals who appear to meet criteria will be invited for a screening visit, when a detailed history and physical exam will be performed by study clinicians. Inclusion and exclusion criteria will be reviewed after the visit to determine study eligibility.

Inclusion criteria:

1. Males or females diagnosed with ongoing post-bariatric hypoglycemia with prior episodes of neuroglycopenia, unresponsive to dietary intervention (low glycemic index, controlled carbohydrate portions) and trial of acarbose therapy at the maximally tolerated dose.
2. Age 18-60 years of age, inclusive, at screening.
3. Willingness to provide informed consent and follow all study procedures, including attending all scheduled visits.

Exclusion criteria:

1. Inability to exercise or medical contraindication to exercise;
2. Documented hypoglycemia occurring in the fasting state (> 12 hours fast);
3. Chronic kidney disease stage 4 or 5 (including end-stage renal disease);
4. Hepatic disease, including serum alanine transaminase (ALT) or aspartate transferase (AST) greater than or equal to 3 times the upper limit of normal; hepatic synthetic insufficiency as defined as serum albumin < 3.0 g/dL; or serum bilirubin > 2.0;
5. Congestive heart failure, New York Heart Association (NYHA) class II, III or IV;
6. History of myocardial infarction, unstable angina or revascularization within the past 6 months or 2 or more risk factors for coronary artery disease including diabetes, uncontrolled hypertension, uncontrolled hyperlipidemia, and active tobacco use;
7. History of syncope (unrelated to hypoglycemia) or diagnosed cardiac arrhythmia;
8. Concurrent administration of β-blocker therapy;
9. History of a cerebrovascular accident;
10. Seizure disorder (other than with suspect or documented hypoglycemia);
11. Active treatment with any diabetes medications except for acarbose and miglitol;
12. Active treatment with a somatostatin analogue (both long and short acting) or diazoxide;
13. Active malignancy, except basal cell or squamous cell skin cancers;
14. Personal or family history of pheochromocytoma or disorder with increased risk of pheochromocytoma(MEN 2, neurofibromatosis, or Von Hippel-Lindau disease);
15. Known insulinoma;
16. Major surgical operation within 30 days prior to screening;
17. Hematocrit < 33% (women) or <36% (men);
18. Bleeding disorder, treatment with warfarin, or platelet count <50,000;
19. Blood donation (1 pint of whole blood) within the past 2 months;
20. Active alcohol abuse or substance abuse;
21. Current administration of oral or parenteral corticosteroids;
22. Pregnancy and/ or Lactation: For women of childbearing potential: there is a requirement for a negative urine pregnancy test and for agreement to use contraception during the study and for at least 1 month after participating in the study. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an intra-uterine device (IUD), the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence;
23. Use of an investigational drug within 30 days prior to screening.

There will be no involvement of special vulnerable populations such as fetuses, neonates, pregnant women, children, prisoners, institutionalized or incarcerated individuals, or others who may be considered vulnerable populations.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Plasma glucose levels in response to physical activity | Blood samples will be collected for measurement of plasma glucose at baseline (pre-exercise), 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, and 180 minutes.
  Area under the curve for glucose levels will be analyzed. Plasma glucose will be measured at baseline, during and after physical activity.
Insulin levels in response to physical activity | Insulin levels are measured at baseline (pre-exercise), 15, 30, 45, 60, 90 and 120 minutes, as well as at the time of hypoglycemia (up to the 120 minute time point, should it occur).
  Area under the curve for insulin levels will be analyzed. Insulin levels will be measured in venous blood obtained through the intravenous catheter.
Glucagon levels in response to physical activity | Glucagon levels are measured at baseline (pre-exercise), 15, 30, 45, 60, 90 and 120 minutes, as well as at the time of hypoglycemia (up to the 120 minute timepoint should it occur).
  Area under the curve for glucagon levels will be analyzed. Glucagon levels will be measured in venous blood obtained through the intravenous catheter.
Glucagon like peptide-1 (GLP-1) levels in response to physical activity | GLP-1 levels are measured at baseline (pre-exercise), 15, 30, 45, 60, 90 and 120 minutes, as well as at the time of hypoglycemia (up to the 120 time point should it occur).
  Area under the curve for GLP-1 levels will be analyzed. GLP-1 levels will be measured in venous blood obtained through the intravenous catheter.

SECONDARY OUTCOMES:
Number of participants who develop hypoglycemia in response to physical activity | Baseline (pre-exercise), assessed up to 180 minutes after the initiation of physical activity.
  Participant displays or reports symptoms of clinically significant hypoglycemia (neuroglycopenia or a venous glucose level of less than 54 mg/dL).
Heart rate variability | Measured once at baseline
  Comparison of R-R interval in milliseconds to normative values
Hypoglycemia symptom score using the Edinburgh Hypoglycemia Symptom Scale (EHSS) | At 60 minute time point, or termination of physical activity if earlier.
  The total EHSS score will be compared between participants. The EHSS total score range is from 18 (which signifies no symptoms of hypoglycemia are present) to 126 (which signifies that the participant has all of assessed for symptoms qualified as very severe). Thus a higher score indicates the presence of both a higher number and/or greater severity of symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States